CLINICAL TRIAL: NCT04861792
Title: The Michigan Sustained Patient-centered Alcohol-Related Care (MI-SPARC) Trial
Brief Title: Michigan SPARC Trial
Acronym: MI-SPARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) - Funder (Unknown); Altarum Institute (Unknown); NORC at the University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: R18HS027076 (AHRQ)
Record Dates: First submitted 2021-04-21; First posted 2021-04-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Alcohol; Drinking; Alcohol Use Disorder (AUD)
Keywords: Alcohol misuse; Unhealthy alcohol use; Alcoholism; Alcohol dependence; Alcohol abuse; Risky drinking
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Originally the SPARC trial was a stepped-wedge cluster-randomized design to evaluate the Michigan SPARC quality improvement intervention compared to usual care. We converted the trial into a program evaluation due to COVID making randomization impossible (e.g., a randomly assigned, unpredictable time to implement was unacceptable in a pandemic, COVID markedly limited primary care practices interest in the trial, and some practices that enrolled closed during the project). The originally planned random assignment to receive the AUD decision aid was not possible due to the small number of participating practices during the pandemic and the need to provide all sites the decision aid to maximize engagement in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients seen before the intervention launch date.
- Quality Improvement Intervention (Experimental): Patients seen after the intervention launch date.
  Interventions: Behavioral: Michigan SPARC Quality Improvement Intervention

INTERVENTIONS:
Behavioral: Michigan SPARC Quality Improvement Intervention — Practice facilitation, electronic health record (EHR) support, performance monitoring and feedback combined with alcohol-related continuing medical education (CME) and maintenance of certification (MOC) and tools to support alcohol related care including a decision aid for shared decision making about alcohol use disorder (AUD).
  Arms: Quality Improvement Intervention

SUMMARY:
Unhealthy alcohol use is a major contributor to morbidity and mortality in the US. Although effective prevention for unhealthy alcohol use and medication treatment for alcohol use disorders (AUDs) can be provided in primary care (PC), they have historically not been included in routine services. As a result, most patients do not receive evidence-based prevention or treatment for unhealthy alcohol use. Several efforts have successfully implemented alcohol-related preventive care-referred to as screening and brief intervention (SBI), but efforts to increase treatment of AUDs with medications have been less successful. Moreover, implementation efforts have usually neglected smaller PC practices, in which most PC is provided.

The Michigan SPARC trial is a partnership between Kaiser Permanente Washington Health Research Institute (KPWHRI) in Seattle, bringing extensive expertise implementing evidence-based alcohol-related care, and Altarum Institute in Ann Arbor, Michigan, bringing demonstrated success engaging over 500 small to medium Michigan-based PC practices in effective quality improvement (QI) efforts. The project builds on Altarum's innovative approach to implementing new or improved clinical care using practice facilitators to provide continuing medical education and maintenance of certification (CME/MOC) programs to PC providers, along with ongoing support for QI using evidence-based implementation strategies. The KPWHRI team recently finished the highly successful AHRQ-funded Sustained Patient-centered Alcohol-Related Care (SPARC) trial using similar implementation strategies in KP Washington, including use of electronic health records and performance monitoring and feedback, and also developed a patient decision aid to support shared decision-making between patients with high-risk drinking and/or AUDs and their PC providers.

The Michigan SPARC trial combines Altarum's expertise in QI in small-medium PC practices in Michigan with KPWHRI's expertise implementing evidence-based prevention and treatment of unhealthy alcohol use-specifically alcohol SBI and medication treatment for AUDs.

Specific Aims of the Michigan SPARC trial had to be markedly modified due to the trial beginning in March 2020 at the same time as the COVID pandemic. A trial was not possible. The revised aims were to describe alcohol screening, brief intervention, AUD diagnosis and initiation of medication treatment for AUD, before and after the Michigan SPARC model was implemented, in small to medium PC practices in Michigan.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years and older
* Seen in primary care at a study practice during the practice's study period

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9590 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Prevention - Screening and brief intervention | For Aim 1 the period up to 6 months before the launch date will be compared to the 6 month period after the launch date.
  The proportion of PC patients who screen positive for unhealthy alcohol use and have BI documented in their EHR.
Treatment - Prescription of AUD medications | For Aim 1 the period up to 6 months before the launch date will be compared to the 6 month period after the launch date.
  The proportion of PC patients who are diagnosed with AUD at a visit who also receive a prescription for medications to treat AUD and are seen for follow-up within 14 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Altarum Institute, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared in the following ways:
  External Evaluator. The Michigan SPARC investigators are committed to working with AHRQ's external evaluator (NORC) on the cross-grant evaluation.
  Other data sharing. We will also make de-identified data available, upon request, after Michigan SPARC trial results are completed and published. No PC practices will be identified in the dataset. Data will be available to investigators who propose a cogent analysis not already part of planned secondary analyses. Proposals must include a biosketch of the Investigator(s), as well as research question(s), sample, measures, methods and statistical issues. Proposals will be reviewed by the Multiple PIs and the leaders of the Michigan SPARC Data and Evaluation team. For approved projects, a data sharing agreement will be developed and subsequently data will be made available.